CLINICAL TRIAL: NCT00843960
Title: Medication Adherence Enhancement in Heart Transplant Recipients: a Randomized Clinical Trial
Brief Title: Medication Adherence Enhancement in Heart Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Dr. rer. biol. hum. Christiane Kugler, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IFB-P46-377
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Medication Adherence; Self Management; Rejection
MeSH Terms: conditions — Medication Adherence; Rejection, Psychology | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): intervention group
  Interventions: Behavioral: behavioral adaptation and symptom management
- 2 (No Intervention): control group

INTERVENTIONS:
Behavioral: behavioral adaptation and symptom management — behavioral adaptation and symptom management
  Arms: 1

SUMMARY:
Medication-related non-adherence increases the risk of rejections and associated graft loss after solid organ transplantation. A randomized controlled intervention will use adherence enhancing strategies out of a larger sample of 300 heart transplant recipients. Non-Adherence will be assessed by patients' self-report and based on immunosuppression level. All non-adherent patients will be randomly designed to either intervention or control group. Multi-module interventions include patient education, electronic medication event monitoring, and a combined behavior and symptom management. Longitudinal follow-up is envisioned after initial intervention.

ELIGIBILITY:
Inclusion Criteria:

* all eligible patients with follow-up at our outpatient clinic
* written informed consent
* sufficient German language skills to read and answer a battery of questionnaires
* > 18 years
* minimum 6 mts post HTX

Exclusion Criteria:

* illiteracy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (composite endpoint) | at month 60

SECONDARY OUTCOMES:
Adherence behavior measurement variables from MEMS system | first 3 month
Immunosuppression level | Month 3, 12 and 60
All individual components of the composite endpoint occurence of adverse events | at month 60
Immunosuppression level | month 12
Immunosuppression level | at month 60

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Kugler, PhD, Principal Investigator — Clinic for Cardiac, Thoracic, Transplantation and Vascular Surgery
Locations (1):
- Clinic for Cardiac, Thoracic, Transplantation and Vascular Surgery, Hanover, Germany

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829